CLINICAL TRIAL: NCT07402044
Title: CAbotégravir LENacapavir DUal Long Acting). Immuno-virological Monitoring and Safety Assessment of HIV-1 Infected Patients Receiving a Long-Acting Antiretroviral Combination of Cabotegravir and Lenacapavir
Brief Title: CABOTEGRAVIR/LENACAPAVIR DUAL LONG ACTING THERAPY (COHORT IMEA 074)
Status: Not yet recruiting | Type: Observational
Sponsor: Institut de Médecine et d'Epidémiologie Appliquée - Fondation Internationale Léon M'Ba (Other)
Collaborators: INSERM UMR S 1136 (Other); ANRS, Emerging Infectious Diseases (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2025-A02118-41; IDRCB (Other: National Agency for Medicines and Health Products Safety.)
Record Dates: First submitted 2025-12-18; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: CABOTEGRAVIR; LENACAPAVIR
Keywords: Lenacapavir; Cabotegravir; HIV; Multicentre cohort

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 48 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The main objective of this national study is to evaluate the virological success of long-acting antiretroviral therapy combining cabotegravir and lenacapavir. The study involves patients who have been receiving this treatment for one year or those for whom the physician decides to initiate it. It also aims to evaluate the tolerability of the treatment and changes in the participants' immunovirological profile during follow-up.

DETAILED DESCRIPTION:
The CALENDULA cohort is a French multicenter study of people living with HIV (PLHIV) receiving long-acting dual therapy combining cabotegravir and lenacapavir (CAB/LEN) for at least 48 weeks.

The study has two parts:

Retrospective part: includes patients who started treatment between July 2024 and the date of the last available follow-up.

Prospective part: includes patients for whom the decision to initiate treatment is made during a 12-month recruitment period, with 48 weeks of follow-up.

No specific intervention is planned; data are simply collected from medical records.

Information will be collected at the following times after the start of treatment:

D0, W24, and W48.

The primary objective is to describe the virological response and tolerance of CAB/LEN dual therapy over 48 weeks.

Virological success is defined as maintaining a viral load (VL) < 50 copies/mL or suppression of VL at W48 without interruption of treatment.

The efficacy criterion is the virological failure rate at S48. The study aims to evaluate the feasibility and tolerability of this innovative therapeutic combination in order to prepare for a future larger-scale study on cabotegravir/lenacapavir.

ELIGIBILITY:
* Age ≥18 years
* HIV-1 infection
* Patients who started taking cabotegravir combined with lenacapavir between July 2024 and the one-year follow-up, or who are due to start taking the CAB/LEN combination.
* Patients who are due to start the CAB/LEN combination following a medical decision.

Exclusion Criteria:

* Participants' objection to the use of follow-up data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: people living with HIV (PLHIV) in France, receiving long-acting dual therapy with cabotegravir/lenacapavir for at least 48 weeks, comprising: (i) a retrospective component, including patients who started this treatment from July 2024 until the last available follow-up data collection; (ii) a prospective component, including patients for whom a medical decision to initiate this treatment is made during a 12-month recruitment period, with a planned follow-up of 48 weeks.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2028-02-15 (Estimated); Study Completion 2028-02-15 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants with virological failure | Week 48
  Two consecutive viral load (VL) measurements ≥50 copies/mL after having achieved VL <50 copies/mL
Percentage of participants with virological failure | Week 24
  ii. A single VL ≥50 copies/mL followed by permanent treatment discontinuation or loss to follow-up after previously achieving VL <50 copies/mL; or discontinuation with VL ≥50 copies/mL
Percentage of participants with virological failure | Week48
  A VL ≥50 copies/mL

SECONDARY OUTCOMES:
1. Percentage of participants with therapeutic success using the FDA Snapshot approach (defined as absence of virological failure, permanent treatment discontinuation, or loss to follow-up). | Week48
2. Percentage of participants with viruses showing resistance-associated mutations. | Week 48
3. Percentage of participants experiencing at least one "blip" | from Week 24 to week 48
4. Plasma concentrations of antiretroviral drugs | from Week 24 to week 48
5. Changes in CD4 and CD8 T-cell counts and in the CD4/CD8 ratio | from enrollment to the end of treatment at 48 weeks
6. Incidence of adverse events and biological abnormalities | from enrollment to the end of the treatment at week 48
7. Changes in body weight and BMI | from the enrollment to the end the treatment at week 48
8. Changes in metabolic parameters | From the enrollment to the end of treatment at week 48
  Total cholesterol, HDL, LDL, Triglycerid, Glyceamia

OTHER OUTCOMES:
3. Percentage of participants experiencing at least one "blip | Week 24
Percentage of participants experiencing at least one "blip | Week 48

CONTACTS AND LOCATIONS:
Overall Officials: Roland LANDMAN, Principal Investigator — Institut de Médecine et d'Epidémiologie Appliquée - Fondation Internationale Léon M'Ba
Locations (13):
- France (13):
  - Victor Dupuy Hospital, Argenteuil
  - Pellegrin Hospital, Bordeaux
  - Saint André Hospital, Bordeaux
  - Raymond poincaré Hospital, Garches
  - Franco-British Hospital (Fbh), Levallois-Perret
  - Hotel Dieu Hospital, Nantes
  - Archet 1Hospital, Nice
  - Bichat Claude Bernard Hospital, Paris
  - Hotel Dieu Hospital, Paris
  - Necker Hospital, Paris
  - Pitié Salpêtrière Hospital, Paris
  - Saint Antoine Hospital, Paris
  - Tourcoing Hospital, Tourcoing

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF